CLINICAL TRIAL: NCT00851903
Title: Combination Therapy of Insulin Glargine and Sitagliptin in Patients With Type 2 Diabetes Not Adequately Controlled by a Previous Treatment With Metformin and Either Insulin Glargine or Sitagliptin
Brief Title: Evaluation of Insulin Glargine in Combination With Sitagliptin in Type 2 Diabetes Patients: EASIE Extension Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXT_LANTU_C_02761; 2008-000521-19 (EudraCT Number)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Sitagliptin Phosphate; Metformin

ARMS (1):
- Combination insulin glargine and sitagliptin (Experimental): Insulin glargine administered once a day, in the evening, at dinner or at bedtime. Starting dose: - last dose administered in the core study for patients previously treated with insulin glargine, - 0.2 U/Kg of body weight for patients previously treated with sitagliptin. Monitoring of blood glucose and titration: all patients, irrespective of their previous treatment group in the core study were empowered to adjust their insulin doses, under strict investigator's supervision. The goal was to achieve through a force titration 70 < Fasting Plasma Glucose (FPG) ≤ 100 mg/dL (3.9 <FPG ≤ 5.5 mmol/L).
  Sitagliptin: stable dose of 100 mg once a day administered with or without food.
  Interventions: Drug: Insulin Glargine; Drug: Sitagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Insulin Glargine — Subcutaneous injection. 100 Units/mL solution for injection in a prefilled SoloStar® pen (3 mL).
  Other Names: Lantus®
Drug: Sitagliptin — Oral administration. 100mg film-coated tablets.
  Other Names: Januvia®
Drug: Metformin — Patients continued with metformin as usual oral anti-diabetic treatment.

SUMMARY:
This study was the extension of the LANTU_C_02761 study named EASIE and identified as NCT00751114 (core study comparing insulin glargine versus sitagliptin in insulin-naïve patients treated with metformin and not adequately controlled).

All patients with Glycosylated Hemoglobin A1c (HbA1c) ≥ 7% at the end of the core study had the possibility to enter this extension study if they met the other inclusion criteria and did not present with any exclusion criteria.

The visit 14 of the core study (week 24) was the visit 1 (baseline, week 0) of the extension study which consisted of a 12-week treatment period.

The objectives of this extension study were:

* To assess the glycemic control (HbA1c <7%) of a 3-month combination therapy with metformin, insulin glargine and sitagliptin in patients not adequately controlled by a previous treatment with metformin plus either insulin glargine or sitagliptin.
* To assess the effect of insulin glargine in combination with sitagliptin on HbA1c level, fasting plasma glucose, 7-point glucose profile, hypoglycemia occurrence, body weight and overall safety.

ELIGIBILITY:
Inclusion criteria:

* Patients who completed the core study LANTU_C_02761 (NCT00751114) i.e. went through the visit 14 investigation,
* HbA1c >= 7 %,
* Dose of metformin compliant with the inclusion criteria of the core study (i.e. at least 1 g/day), and maintained stable for the duration of the core study
* Ability and willingness to perform plasma blood glucose monitoring using the sponsor-provided plasma glucose meter and to complete the patient dairy,
* Signed informed consent obtained prior any study procedure,
* Willingness and ability to comply with the study protocol.

Exclusion Criteria:

* Treatment with oral antidiabetic drugs other than metformin and sitagliptin in the core study,
* Treatment with insulin other than Insulin Glargine in the core study (except in case of an emergency, for a period of time less than 7 days),
* Treatment with a non-permitted drug during the core study,
* Pregnant or lactating women,
* In-patient care,
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study (an optic fundus examination should have been performed within the 2 years prior to study entry in the core study),
* Impaired renal function: serum creatinine >= 1.5 mg/dL (>= 133µmol/L) or >= 1.4 mg/dL (>=124 µmol/L) in men and women, respectively,
* History of sensitivity to the study drugs or to drugs with a similar chemical structure,
* Impaired hepatic function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 3 x upper limit of normal range,
* Alcohol or drug abuse within the last year,
* Night shift worker,
* Presence of any condition (medical, psychological, social or geographical), current or anticipated that the investigator feels would compromise the patient's safety or limit the patient successful participation in the study,
* Treatment with weight loss medications (e.g. sibutramine, orlistat, rimonabant),
* History of pancreatitis.

Ages: 35 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Kallithea, Greece
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Beirut, Lebanon
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 445 patients who completed the EASIE study, 194 had an endpoint Glycosylated Hemoglobin A1c (HbA1c) ≥ 7%. A total of 112 patients were included in the extension study: 37 uncontrolled on previous treatment with metformin and insulin glargine and 75 uncontrolled on previous treatment with metformin and sitagliptin in the EASIE study.
Pre-assignment Details: Among the 112 included patients, two patients prematurely discontinued from the study. One of them had continued his sitagliptin treatment but never started the insulin glargine treatment.
Period: Overall Study
Arm/Group | Combination Insulin Glargine and Sitagliptin
Started | 112
Safety Population | 112 (patients treated with at least one dose of insulin glargine OR one dose of sitagliptin)
Treated by Combination | 111 (patients treated with at least one dose of insulin glargine AND one dose of sitagliptin)
Modified Intent-To-Treat Population | 111 (mITT population: patients treated by combination with at least 1 on-treatment efficacy measure)
Completed | 110
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Combination Insulin Glargine and Sitagliptin: Insulin glargine administered once a day, in the evening, at dinner or at bedtime. Starting dose: - last dose administered in the core study for patients previously treated with insulin glargine, - 0.2 U/Kg of body weight for patients previously treated with sitagliptin. Monitoring of blood glucose and titration: all patients, irrespective of their previous treatment group in the core study were empowered to adjust their insulin doses, under strict investigator's supervision. The goal was to achieve through a force titration 70 <FPG ≤ 100 mg/dL (3.9 <FPG ≤ 5.5 mmol/L).
  Sitagliptin: stable dose of 100 mg once a day administered with or without food.
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 111
Age Continuous [Mean (Standard Deviation); unit: years] — mITT population
  Age collected at EASIE study entry (24 weeks before baseline)
  years | 52.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — mITT population
  Participants
    Female | 56
    Male | 55
Body Weight [Mean (Standard Deviation); unit: kg] — mITT population
  kg | 84.6 (21.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — mITT population
  kg/m² | 31.3 (5.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mITT population
  mmHg | 129.9 (15.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — mITT population
  mmHg | 80.1 (7.3)
Heart Rate [Mean (Standard Deviation); unit: beats/min] — mITT population
  beats/min | 76.9 (9.1)
Duration of diabetes [Median (Inter-Quartile Range); unit: years] — mITT population
  Duration of diabetes collected at EASIE study entry (24 weeks before baseline)
  years | 4.1 (5.1) [2.0 to 8.3]
At least one diabetic late complication [Number; unit: participants] — mITT population
  Diabetic late complications: myocardial infarction, angina pectoris, coronary artery disease, heart failure, stroke, transient ischemic attack, peripheral vascular disease, diabetic neuropathy, diabetic nephropathy, diabetic retinopathy
  Information collected at EASIE study entry (24 weeks before baseline)
  participants
    Yes | 23
    No | 88
Glycosylated Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] — mITT population
  percent | 8.0 (1.0)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values N=110
  mg/dL | 151.5 (46.9)
Self-Monitored Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — mITT population but due to missing values N=104
  mg/dL | 144.4 (38.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Response Rate: Percentage of Patients Achieving Glycosylated Haemoglobin A1c (HbA1c) < 7% at Study Endpoint (End of Treatment Period)
Time Frame: study endpoint: week 12 or earlier in case of premature discontinuation
Population: The population analyzed consisted of the subset of mITT patients who had HbA1c value at study endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 106
percentage of participants | 51.9 [41.97 to 61.70]

2. Secondary Outcome: HbA1c: Change From Baseline to Study Endpoint
Description: Change = study endpoint - baseline
Time Frame: baseline, study endpoint: week 12 or earlier in case of premature discontinuation
Population: The population analyzed consisted of the subset of mITT patients who had both baseline and endpoint for this outcome measure
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 106
percent | -0.80 (1.05)

3. Secondary Outcome: Self-Monitored Fasting Plasma Glucose (SMFPG) Mean : Change From Baseline to Study Endpoint
Description: SMFPG mean = mean of the fasting plasma glucose values recorded on the 6 consecutive days before the visit (at least 3 values needed).
  Change = study endpoint - baseline.
Time Frame: baseline, study endpoint: week 12 or week 8 if value not available at week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 104
mg/dL | -35.43 (39.61)

4. Secondary Outcome: 7-point Plasma Glucose Profile: Change From Baseline to Study Endpoint
Description: 7-point plasma glucose recorded before and after breakfast, before and after lunch, before and after dinner and at bedtime.
  Change = study endpoint - baseline.
Time Frame: baseline, study endpoint: week 12 or week 8 if value not available at week 12
Population: The population analyzed consisted of the subset of mITT patients who had valid 7-point plasma glucose profiles (4 points needed for a valid profile) both at baseline and endpoint.
  Depending on the time point, few values were missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 104
mg/dL
  Before breakfast (N=104) | -34.2 (38.1)
  After breakfast (N=103) | -34.1 (48.1)
  Before lunch (N=104) | -26.6 (48.2)
  After lunch (N=104) | -26.5 (43.7)
  Before dinner (N=103) | -25.1 (43.0)
  After dinner (N=100) | -24.9 (46.7)
  At bedtime (N=93) | -35.2 (51.7)

5. Secondary Outcome: Insulin Dose
Description: Daily dose at the face-to-face visits
Time Frame: baseline, week 4, week 8, week 12
Population: mITT population
Measure: Mean (Standard Deviation); unit: unit per kg body weight
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 111
unit per kg body weight
  Baseline | 0.28 (0.18)
  Week 4 N=110 | 0.37 (0.16)
  Week 8 N=110 | 0.42 (0.18)
  Week 12 | 0.46 (0.20)

6. Secondary Outcome: Number of Patients With at Least One Episode of Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was defined as an event with clinical symptoms that were considered to result from hypoglycemia confirmed or not by a plasma glucose measurement <= 70mg/dL [3.9 mmol/L]
Time Frame: During the treatment period (12 weeks) plus 7 days after last dose
Population: The population analyzed for this outcome measure was the safety population
Measure: Number; unit: participants
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 112
participants | 40

7. Secondary Outcome: Change in Body Weight From Baseline to Study Endpoint
Description: Change = study endpoint - baseline
Time Frame: baseline, study endpoint: week 12 or week 8 or week 4 depending on last available value
Population: The population analyzed was the safety population with both baseline and endpoint values available
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Combination Insulin Glargine and Sitagliptin
Number analyzed (Participants) | 111
kg | 1.15 (2.24)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the extension study (12 weeks). Only adverse events starting from inclusion in the extension study were taken into account.
Arm/Group | Combination Insulin Glargine and Sitagliptin
Serious Adverse Events (participants affected / at risk) | 2/112
Other Adverse Events (participants affected / at risk) | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Insulin Glargine and Sitagliptin (N=112)
Right ventricular failure (Cardiac disorders) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 45 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.